CLINICAL TRIAL: NCT01929057
Title: Evaluation of the Role of Propionibacterium Acnes in the Inflammatory Lesions Associated With Acne Vulgaris
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tissa Hata, MD, MD, University of California, San Diego
Other Study IDs: 121230
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acne patients: This group consists of patients who have at least moderate to severe acne on their back
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw
- Healthy Controls: This group contains participants who do not have any active acne lesions on their back
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw

INTERVENTIONS:
Procedure: Skin biopsy — 4-millimeter punch biopsies will be performed on all subjects (acne patients and healthy controls)
Procedure: Blood draw — Approximately half a tube of blood will be drawn from all participants in the study

SUMMARY:
The purpose of this study is to determine the response of acne patients and healthy control patients to the P. acnes bacteria. Half a tube of blood will be drawn from all participants to determine whether or not they have antibodies to the P. acnes bacterium. Anywhere from 1 to 4 skin biopsies of acne pimples or normal control skin will be taken from all subjects for further analysis in the lab to determine whether the inflammation in these pimples can be reduced using anti-P.acnes antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Fits into one of the following diagnostic groups:

  1. Healthy subject with no active skin disease or history of skin disease
  2. Diagnosis of moderate-to-severe truncal acne diagnosed clinically and confirmed using the modified Leeds criteria with no reported use of topical acne treatments within the past 2 weeks prior to enrollment in the study, and no reported use of oral acne treatments during the past 4 weeks prior to enrollment in the study
  3. Diagnosis of moderate-to-severe truncal acne diagnosed clinically and confirmed using the modified Leeds criteria who has used any topical acne treatments in the 2 weeks prior to enrolling in the study, or who has used any oral acne treatments during the 4 weeks prior to enrolling in the study 2. Age 18-60 years 3. Male or female of any race and ethnicity 4. Subject agrees to comply with study requirements

Exclusion Criteria:

1. Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study
2. Subject has Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
3. Pregnant or nursing females
4. Immunocompromised subjects (e.g., lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome), or with a history of active or malignant disease (excluding non-melanoma skin cancer) as determined by the participant's medical history.
5. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
6. Subjects with significant concurrent medical condition(s) at screening that in the view of the investigator prohibits participation in the study (e.g., severe concurrent allergic disease, condition associated with malignancy, and condition associated with immunosuppression)
7. Active viral or fungal skin infections at the target areas
8. Are currently receiving lithium now or within the last 4 weeks.
9. Ongoing participation in an investigational drug trial
10. Use of any systemic immunosuppressive therapy less than four weeks prior to screening.
11. Subjects with diabetes
12. Injured, broken skin that, per the investigator, may lead to poor wound healing
13. Subjects with allergies to anesthetic medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tissa Hata, MD, Principal Investigator — UCSD
Locations (1):
- UCSD Division of Dermatology, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acne Patients | Healthy Controls
Started | 31 | 3
Completed | 31 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acne Patients | Healthy Controls | Total
Number analyzed (Participants) | 31 | 3 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (6.7) | 26 (2.3) | 26 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 2 | 19
  Male | 14 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 25 | 3 | 28
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 3 | 34

OUTCOME MEASURES:

1. Primary Outcome: Level of IL-1β
Description: The amount of IL-1β, an inflammatory marker, is measured in skin biopsies obtained from healthy patients and compared with levels in biopsies of acne lesions.
Time Frame: post biopsy
Measure: Mean (Standard Deviation); unit: pg/mg
Units Other Than Participants: Biopsies
Arm/Group | Healthy Controls | Acne Patients
Number analyzed (Participants) | 3 | 31
Number analyzed (Biopsies) | 3 | 31
pg/mg | 52.5 (15.6) | 361.2 (60.3)

2. Secondary Outcome: Level of Antibody to CAMP(Christie-Atkins-Munch-Petersen) Factor
Description: Antibody titers were determined by using recombinant CAMP factor or green fluorescent protein (GFP) as a capture antigen for coating onto a enzyme-linked immunosorbent assay (ELISA) plate. The endpoint was defined as the dilution of serum on CAMP factor-coated wells producing the same Optical Density(570-450) as a 1/100 dilution of serum on GFP-coated wells. Sera negative at the lowest dilution tested were assigned endpoint titers of 100. The data were presented as geometric mean endpoint ELISA titers.
Time Frame: post biopsy
Measure: Geometric Mean (Standard Error); unit: titers
Arm/Group | Acne Patients | Healthy Controls
Number analyzed (Participants) | 31 | 3
titers | 280 (99) | 625 (122)

ADVERSE EVENTS:
Arm/Group | Acne Patients | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/3
Other Adverse Events (participants affected / at risk) | 0/31 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No